CLINICAL TRIAL: NCT01967121
Title: Compex Use With Delayed Onset Muscle Soreness: A Comparison to Other Methods
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michigan State University (Other)
Responsible Party: Principal Investigator, Tracey Covassin, Associate Professor, Michigan State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB# 13-849F
Record Dates: First submitted 2013-10-16; First posted 2013-10-22 (Estimated); Results first posted 2014-08-29 (Estimated); Last update posted 2014-08-29 (Estimated); Status verified 2014-08

CONDITIONS: Focus of Study is to Determine Efficacy of Compex
Keywords: Compex, ice

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 'Compex unit's Active Recovery® program' (Experimental): The Compex electrical stimulation system utilized in this study is intended for external application with electrodes to create a muscular contraction and help enhance recovery after eccentric muscular activity.
  Interventions: Device: Compex unit's Active Recovery® program
- Ice application (Other): A randomized pre and post-test research design will be used to compare three interventions (control, ice, compex) to alleviate the physical symptoms of delayed-onset muscle soreness (DOMS).
  Interventions: Other: Ice application
- Control (No Intervention): This is a control group where subjects will not perform an intervention.

INTERVENTIONS:
Device: Compex unit's Active Recovery® program — Compex unit's Active Recovery® program will be performed for 15 minutes once per day.
  Arms: 'Compex unit's Active Recovery® program'
Other: Ice application — Participants will apply ice on their hamstring for 15 minutes three times per day until muscle soreness is no longer present
  Arms: Ice application

SUMMARY:
The purpose of this research study is to determine if the application of ice, control group, or a muscle stimulation program from the Compex® series can help reduce or eliminate delayed muscle soreness from performing leg extension and flexion. Individuals will complete a health history questionnaire to determine if they qualify for this study. We will measure your leg girth with a measuring tape and take a pain measurement of your hamstrings by using a spring to press down on your leg. Individuals will then warm-up on a bike without resistance for 5 minutes followed by 10 regular leg extension and flexion exercises. Individuals will then perform 6 sets of 10 leg extension and flexion exercises on a biodex machine (similar to leg curl machines in the gym). Individuals will perform each set to the maximum effort of their capables. After each set of 10 individuals will have a 2 minute rest. We will ask you to rank your leg soreness on a scale from 1-10.

Individuals will then be assigned to a modality of either ice, control group or compex. Individuals will perform the modality (ice, control, compex) we assign you to until you are no longer sore.

Over the next five days individuals will return to measure their level of soreness, leg girth and pain pressure.

This study will examine the following hypotheses:

H1: There will be no difference in pressure pain threshold after using the Compex compared to other groups.

H2: There will be no difference in perceived soreness after using the Compex compared to other groups.

H3: There will be no difference in muscular strength after using the Compex compared to other groups.

H4: There will be no difference in active range of motion after using the Compex compared to other groups.

ELIGIBILITY:
Inclusion Criteria:

* The studied population will be composed of 45 physically active college students between the ages of 18-30 years old.
* Inclusionary criteria will be participation in a physical activity as defined by the ACSM, which can be a mixture of moderate (i.e., sufficient to raise the heart rate and begin to sweat) and vigorous (i.e., breathing hard and fast with a rapidly rising heart rate) intensity aerobic activity and muscle strengthening (i.e., weights lifted to the point where anther repetition cannot be completed without help) activities two or more time per week (ACSM, 2011.)

Exclusion Criteria:

* Exclusionary criteria will be surgery within the last six months requiring immobilization for more than four weeks, discomfort performing intense physical activity, diseases like muscular dystrophy that predispose muscular damage beyond reasonable levels resulting from physical activity, and current injury of the knees or hips.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2013-10; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tracey Covassin, PhD, Principal Investigator — Michigan State University
Locations (1):
- Michigan State University, East Lansing, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 'Compex Unit's Active Recovery® Program' | Ice Application | Control
Started | 25 | 25 | 25
Completed | 25 | 25 | 25
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants first had their leg girth measured with a measuring tape. Pain measurement was taken using a syringe with spring in place of algometer six and 12 inches above the popliteal fossa for tenderness. After completing the visual analog scale, participants completed the induction DOMS protocol.
Groups:
- Total: Total of all reporting groups
Arm/Group | 'Compex Unit's Active Recovery® Program' | Ice Application | Control | Total
Number analyzed (Participants) | 25 | 25 | 25 | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.43 (1.25) | 19.61 (1.68) | 19.78 (1.89) | 19.64 (1.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 15 | 45
  Male | 10 | 10 | 10 | 30

OUTCOME MEASURES:

1. Primary Outcome: Pain Scores on the Visual Analog Scale
Description: Visual Analog Scale for Muscle Soreness scale The scale for measuring the intensity of muscle soreness will be a 10 cm visual analog scale, spaced by one centimeter increments from one to 10. Ten will represent the maximum amount of soreness and zero represents no soreness at all. Subjects will be asked to complete this scale once per day at the same time of day until the soreness has dissipated. The Visual Analog Scale for muscle soreness is measured as 'scores on a scale'.
Time Frame: Day 1 through Day 5
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | 'Compex Unit's Active Recovery® Program' | Ice Application | Control
Number analyzed (Participants) | 25 | 25 | 25
scores on a scale
  Day 1 | 2.64 (2.21) | 2.60 (2.81) | 2.45 (2.10)
  Day 2 | .80 (1.5) | .72 (1.24) | .85 (1.5)
  Day 3 | .4 (.82) | .56 (1.23) | .88 (1.72)
  Day 4 | .16 (.55) | .44 (.92) | .70 (1.78)
  DAY 5 | .04 (.2) | .16 (.55) | .4 (1.39)

ADVERSE EVENTS:
Arm/Group | 'Compex Unit's Active Recovery® Program' | Ice Application | Control
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No